CLINICAL TRIAL: NCT01135927
Title: A Trial Investigating the Pharmacodynamic Properties of NN1250 in Japanese Subjects With Type 1 Diabetes
Brief Title: A Trial Investigating the Effect of NN1250 in Japanese Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1250-1996; U1111-1113-6722 (Other: WHO); JapicCTI-101158 (Other: JAPIC)
Record Dates: First submitted 2010-05-31; First posted 2010-06-03 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Detemir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: insulin degludec
- B (Active Comparator)
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin degludec — NN1250 (insulin degludec) injected s.c. (under the skin) once daily for 6 days
  Arms: A
Drug: insulin detemir — Insulin detemir injected s.c. (under the skin) once daily for 6 days
  Arms: B

SUMMARY:
This trial is conducted in Japan. The aim of this clinical trial is to investigate the effect of NN1250 (insulin degludec) in Japanese subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Treated with multiple daily insulin injections or continuous subcutaneous insulin infusion (CSII) for at least 12 months
* Current daily basal insulin requirement above or equal to 0.3 (I)U/kg/day
* Glycosylated haemoglobin A1c (HbA1c) below or equal to 10.0% (one retest within a week is permitted with the result of the last test being conclusive)

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Surgery or trauma with significant blood loss (more than 500 mL) within the last 3 months prior to screening
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)
* Not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period (only clamp period)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Area under the NN1250 GIR (glucose infusion rate) curve | During one dosing interval at steady state

SECONDARY OUTCOMES:
Area under the serum insulin detemir concentration-time curve | During one dosing interval at steady state

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- [Result] Ikushima I, Kaku K, Hirao K, Bardtrum L, Haahr H. Pharmacokinetic and pharmacodynamic properties of insulin degludec in Japanese patients with type 1 diabetes mellitus reflect similarities with Caucasian patients. J Diabetes Investig. 2016 Mar;7(2):270-5. doi: 10.1111/jdi.12399. Epub 2015 Aug 27. PMID 27042281
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com